CLINICAL TRIAL: NCT04749238
Title: Safety and Efficacy Assessment of NucleoCapture Selective DNA Adsorber in Humans
Brief Title: Effect of Extracorporeal Adsorption of Plasma Neutrophil Extracellular Traps (NET) in Sepsis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Santersus AG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Nucleo 514/2020
Record Dates: First submitted 2021-01-28; First posted 2021-02-11 (Actual); Last update posted 2022-12-06 (Actual); Status verified 2022-12

CONDITIONS: Sepsis; Sepsis-associated AKI
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment with NucleoCapture device (Experimental): Device: 100 ml NucleoCapture selective DNA adsorber. Treatment with NucleoCapture in one arm.
  Interventions: Device: NucleoCapture device

INTERVENTIONS:
Device: NucleoCapture device — Device: 100 ml NucleoCapture selective DNA adsorber. Treatment with NucleoCapture in one arm
  Other Names: NucleoCapture selective DNA adsorber

SUMMARY:
This open non-randomized controlled single center study investigates to what extent the removal of circulating Neutrophil Extracellular Traps (NETs) from blood by NucleoCapture device has a positive effect on the treatment of patients with sepsis and sepsis-associated AKI (SA-AKI).

DETAILED DESCRIPTION:
The term "sepsis" refers to a clinical syndrome in which a dysregulation of the host's inflammatory reaction to infection leads to a life-threatening of organ dysfunctions. Sepsis and septic shock are major causes of death in intensive care units worldwide. Sepsis remains the most important cause of AKI in the intensive care unit (ICU) with 15%-20% of patients with sepsis-associated AKI (SA-AKI) prescribed RRT . In addition to association with short term mortality, AKI is also linked to the later development of CKD, ESRD, and long-term increased risk of death

NETosis is a unique form of neutrophil cell death that is characterized by the release of neutrophil extracellular traps (NETs) composed of DNA web-like structures decorated with highly cytotoxic protein components. Release of NETs leads to bystander tissue damage (including the kidneys) and drives a fatal course of disease in sepsis patients.

The plasmapheresis is a medical procedure, where pathogenic components are being removed from the blood by adsorbers outside the body in an extracorporeal circulation. For removal of the pathogenic substances the plasma is separated from the blood to pass the adsorber. The purified plasma is merged with the solid blood components thereafter and returned to the patient. The NucleoCapture device provide highly selective removal of neutrophil extracellular traps from human blood during plasmapheresis procedure.

ELIGIBILITY:
Inclusion Criteria:

* Male or female ≥ 18 and ≤ 75 years of age.
* Meet the clinical criteria of sepsis according to the Third International Consensus Definitions for Sepsis and Septic Shock (Sepsis-3))
* Written informed consent

Exclusion Criteria:

* A terminal state
* Active bleeding or uncontrolled acute massive bleeding

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2021-01-26 (Actual); Primary Completion 2021-10-24 (Actual); Study Completion 2021-10-24 (Actual)

PRIMARY OUTCOMES:
Incidence of acute kidney injury (AKI) | from [start of treatment] through 28 days after
  Incidence of acute kidney injury (AKI) in accordance with Kidney Disease Improving Global Outcomes (KDIGO) definitions for AKI
Severity of acute kidney injury (AKI) | from [start of treatment] through 28 days after
  Severity of acute kidney injury (AKI) in accordance with KDIGO definitions for AKI
Rate of AKI transition to the more severe stage (for patients with AKI at baseline). | from [start of treatment] through 28 days after
  Rate of worsening of acute kidney injury (AKI) in accordance with KDIGO AKI classification (Changing stages from 1 to 2, from 2 to 3).
Serum creatinine change over time | from [start of treatment] through 28 days after
  Change of creatinine in serum over time for each patient and in average in group
Serum urea change over time | from [start of treatment] through 28 days after
  Change of urea in serum over time for each patient and in average in group
Urine output change | from [start of treatment] through 28 days after
  Change of urine output over time for each patient and in average in group

SECONDARY OUTCOMES:
All-cause mortality | from [start of treatment] through 28 days after
  Mortality for any reasons for each patient and in average in group
SOFA scores change | from [start of treatment] through 28 days after
  Change in SOFA scores over time for each patient and in average in group
qSOFA scores change | from [start of treatment] through 28 days after
  Change in qSOFA scores over time for each patient and in average in group

OTHER OUTCOMES:
Blood level of neutrophil extracellular traps (NETs) change over time | from [start of treatment] through 28 days after
  Change of NETs in blood over time for each patient and in average in group

CONTACTS AND LOCATIONS:
Locations (1):
- North-Western Regional Scientific and Clinical Center named after L.G. Sokolov, Saint Petersburg, Russia

IPD SHARING:
Plan to Share IPD: Undecided